CLINICAL TRIAL: NCT06502353
Title: A Pilot Study to Investigate the Use of the Plexaa Preconditioning Device (BLOOM43) for Gender Affirming Mastectomy - a Prospective Cohort Study
Brief Title: Plexaa For Preconditioning: Gender Affirming Mastectomy
Acronym: P4PGAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Plexaa Ltd (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 75139; Pro00074534 (Other: Advarra)
Record Dates: First submitted 2024-06-26; First posted 2024-07-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Nipple Necrosis; Nipple Graft Loss
Keywords: Nipple necrosis; Nipple graft loss; Preconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (single arm) (Experimental): Each patient will be given the device, BLOOM43, for use at home. It will be worn in a patient's existing bra over their right breast and the preconditioning protocol will be done 12 hours before surgery - i.e. the evening before. Patients will then attend their breast surgery the next day as planned.
  Interventions: Device: BLOOM43

INTERVENTIONS:
Device: BLOOM43 — Heat preconditioning
  Other Names: Plexaa preconditioning device

SUMMARY:
The goal of this clinical trial is to evaluate the use of the Plexaa preconditioning device (BLOOM43) in transgender and non-binary patients undergoing gender affirming mastectomy. This study aims to understand a participant's experience of the device, including its usability and acceptability.

Participants will use the device to precondition their right breast the evening before undergoing surgery (gender affirming mastectomy).

ELIGIBILITY:
Inclusion Criteria:

* All transgender or non-binary patients over the age of 18 years (no maximum age limit)
* Patients undergoing peri-areolar mastectomy or double incision mastectomy with a free nipple graft for gender affirmation

Exclusion Criteria:

* Patients undergoing surgery for breast cancer
* Delayed (two-stage) breast reconstruction patients
* Patients undergoing simple mastectomy or wide local excision of a breast tumour
* Presence of open breast skin wounds, or infected or inflamed breast skin
* Presence of a cardiac pacemaker, defibrillator or any other implantable electronic device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Participant experience | 30 days
  Participants' experience of the device will be evaluated with the use of a questionnaire. Most of the questions will consist of multiple-choice components with a five-point scale and there will also be a section for further comments from participants.

SECONDARY OUTCOMES:
Compliance | 1 day
  Proportion of participants who are compliant with the preconditioning protocol
Nipple necrosis/nipple graft loss | 30 days
  Proportion of participants experiencing partial or complete nipple necrosis/nipple graft loss and the rate of hospital readmission due to this

CONTACTS AND LOCATIONS:
Overall Officials: Dung Nguyen, Principal Investigator — Stanford University
Locations (1):
- Division of Plastic & Reconstructive Surgery, Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meerwijk EL, Sevelius JM. Transgender Population Size in the United States: a Meta-Regression of Population-Based Probability Samples. Am J Public Health. 2017 Feb;107(2):e1-e8. doi: 10.2105/AJPH.2016.303578. PMID 28075632
- [Background] Rifkin WJ, Robinson IS, Kloer C, Cripps CN, Boyd CJ, Blasdel G, Zhao LC, Bluebond-Langner R. Gender-affirming Mastectomy: Comparison of Periareolar and Double Incision Patterns. Plast Reconstr Surg Glob Open. 2022 May 25;10(5):e4356. doi: 10.1097/GOX.0000000000004356. eCollection 2022 May. PMID 35646495
- [Background] Perez-Alvarez IM, Zolper EG, Schwitzer J, Fan KL, Del Corral GA. Incidence of Complications in Chest Wall Masculinization for the Obese Female-to-Male Transgender Population: A Case Series. World J Plast Surg. 2021 May;10(2):14-24. doi: 10.29252/wjps.10.2.14. PMID 34307093
- [Background] Kankam HKN, Mehta S, Jain A. Thermal Preconditioning for Surgery: A Systematic Review. J Plast Reconstr Aesthet Surg. 2020 Sep;73(9):1645-1664. doi: 10.1016/j.bjps.2020.05.025. Epub 2020 May 21. PMID 32505626
- [Background] Mehta S, Rolph R, Cornelius V, Harder Y, Farhadi J. Local heat preconditioning in skin sparing mastectomy: a pilot study. J Plast Reconstr Aesthet Surg. 2013 Dec;66(12):1676-82. doi: 10.1016/j.bjps.2013.07.034. Epub 2013 Sep 4. PMID 24011908
- [Background] Mehta S, Cro SC, Coomber B, Rolph R, Cornelius V, Farhadi J. A randomised controlled feasibility trial to evaluate local heat preconditioning on wound healing after reconstructive breast surgery: the preHEAT trial. Pilot Feasibility Stud. 2019 Jan 11;5:5. doi: 10.1186/s40814-019-0392-y. eCollection 2019. PMID 30656059